CLINICAL TRIAL: NCT02602314
Title: Sustained Treatment-free Remission in BCR-ABL+ Chronic Myeloid Leukemia: a Prospective Study Comparing Nilotinib Versus Imatinib With Switch to Nilotinib in Absence of Optimal Response. SUSTRENIM Study - GIMEMA CLM1415
Brief Title: Sustained Treatment-free Remission in BCR-ABL+ Chronic Myeloid Leukemia
Acronym: SUSTRENIM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CML1415
Record Dates: First submitted 2015-11-10; First posted 2015-11-11 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Chronyc Myeloid Leukemia
Keywords: Chronic myeloid leukemia; Nilotinib; Imatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Imatinib + Nilotinib (Experimental)
  Interventions: Drug: Imatinib; Drug: Nilotinib
- Nilotinib (Experimental)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Imatinib
  Arms: Imatinib + Nilotinib
Drug: Nilotinib

SUMMARY:
The study will investigate in newly diagnosed CP-CML patients the efficacy of NIL frontline therapy vs IM followed by switch to NIL in the case of absence of optimal response as defined by the ELN criteria.

DETAILED DESCRIPTION:
This is a prospective, interventional, randomized, two arms, phase IV study evaluating both the depth of the molecular response and the rate of treatment free remission rate in newly diagnosed CP-CML patients treated with NIL or IM followed by switch to NIL in absence of optimal response (defined according the ELN 2013 criteria) as per clinical practice.

The enrolled patients will be randomized 1:1 between NIL and IM. Patients will be stratified according to the Sokal risk score to high versus intermediate/low risk groups. Newly diagnosed patients will be treated according to the registered dose of NIL and IM for frontline chronic phase CML (300 mg BID and 400 mg OAD, respectively). The patients intolerant to IM and the patients without optimal response to IM at 3 months, at 6 months, at 12 months (except the patients with progression to accelerated or blastic phase) will be switched to NIL second line.

The absence of optimal response is defined by at least one of the following ELN criteria: a) Absence of Complete Hematologic Response at 3 months or thereafter; b) Absence of Partial Cytogenetic Response (> 35% Ph+ metaphases) at 3 months; c) BCR-ABL transcript level > 10% according to the IS at 3 months; d) Absence of Complete Cytogenetic Response (> 1% Ph+ metaphases) at 6 months; e) BCR-ABL transcript level > 1% according to the IS at 6 months; f) Absence of Major Molecular Response (MR3.0, transcript level > 0.1% according to the IS) at 12 months.

Treatment choice for the patients with progression to advanced disease phase while on IM and for the patients intolerant to or resistant (including progressions to advanced phases) to NIL will be up to the principal investigator of the participating Center. However, information concerning the course and outcome of these patients will be collected and recorded for at least 5 years, and they could be enrolled in investigational studies promoted by GIMEMA or other sponsors.

After the induction of deep molecular remission phase of therapy, i.e. the first two years of the study, residual disease will be closely monitored (quarterly) by Q-PCR assays. All the patients who obtain a reduction greater than 4.0 logs of residual disease (MR4.0) within the first three years of treatment, and maintain this level of response in all the subsequent tests up to the end of the fourth years of therapy qualify for the discontinuation phase of the study. Therefore, all patients who are in MR4.0 after a four-year period of TKI treatment, that must include in its final part at least one years of maintained MR4.0, defined as 12-month period during which the MR4.0 never is lost in 4 consecutive MRD analyses at three-monthly intervals, will enter the treatment free remission (TFR) phase of the study. In case of loss of MR3.0, the last assumed TKI will be resumed at the same dose.

All patients, including those who do not match the criteria for discontinuation of TKI treatment, will continue the assigned treatment and will be followed for 5 years, starting from the date of enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of BCR/ABL+ CML in chronic phase

Documented chronic phase CML must meet all the following criteria:

< 15% blasts in peripheral blood < 30% blasts plus promyelocytes in peripheral blood < 20% basophils in the peripheral blood

* 100 x 109/L (≥ 100,000/mm3) platelets

  * Age ≥18
  * ECOG performance status of 0-2
  * Evidence of typical BCR-ABL transcripts which are amenable to standardized RQ-PCR
  * Adequate end organ function as defined by:

Total bilirubin < 1.5 x ULN (ULN = upper limit of normal in a local institution lab).

Does not apply to patients with isolated hyperbilirubinemia (e.g., Gilbert's disease) grade < 3 SGOT (AST) and SGPT (ALT) ≤ 3 x ULN Serum amylase and lipase ≤ 2 x ULN Alkaline phosphatase ≤ 2.5 x ULN Serum creatinine < 1.5 x ULN

* Having completed the QoL baseline evaluation (i.e., before randomization)
* Written informed consent prior to any study procedures.

Exclusion Criteria:

* Expression of any atypical BCR-ABL transcripts, instead of the classical P210-encoding type with the e13a2 or the e14a2 junction at screening.
* Previous treatment with BCR-ABL inhibitors for a period longer than 1 month.
* Previous anticancer agents (hydroxyurea, anagrelide, interferon) for CML for a time longer than three months.
* Poorly controlled diabetes mellitus (defined as HbA1c >8%).
* Prior documented history of coronary heart disease, including myocardial infarction, coronary bypass, coronary stent, and symptomatic angina:

LVEF <45% or below the institutional lower limit of the normal range (whichever ishigher) Complete left bundle branch block Right bundle branch block plus left anterior or posterior hemiblock Use of a ventricular-paced pacemaker Congenital long QT syndrome or a known family history of long QT syndrome History of or presence of clinically significant ventricular or atrial tachyarrhythmias

* Atrial fibrillation or flutter
* Clinically significant resting bradycardia (< 50 beats per minute)
* QTc > 450 msec on the average of three serial screening ECGs (using the QTcF formula). If QTcF > 450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and the patient re-tested History or clinical signs of myocardial infarction within 12 months of study entry History of unstable angina within 12 months of study entry Other clinically significant heart disease (e.g. congestive heart failure)

  * Uncontrolled hypertension is not a heart disease.
  * History of peripheral arterial occlusive disease.
  * History of acute pancreatitis within 12 months of study entry, or a past medical history of chronic pancreatitis.
  * Patients actively receiving therapy with strong CYP3A4 inhibitors and/or inducers which cannot be either discontinued or switched to a different medication prior to starting study drug.
  * Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and for which cannot be either safely discontinued or switched to a different medication prior to starting study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Number of of patients with molecular response | At 24 months from study entry
Number of patients who remain in sustained treatment free remission, without molecular relapse | After 12 months after entering the treatment-free-remission (TFR) phase

SECONDARY OUTCOMES:
Number of patients with molecular response | 4 years after study entry
Number of patiens in progression-free survival | 5 years after study entry
Number of patients with major molecular response | At 1, 2, 3 and 4 years from study entry
Number of toxic events | At 5 years from study entry
Number of patients who discontinue treatment | At 5 years from study entry
Number of patients with quality of life differences between treatment arms over time | At baseline and at 3, 6, 12, 18, 24, 30, 36, 42, 48, and 60 months from study entry.
  To assess the patient-reported quality of life (QoL) and adherence to therapy at baseline and at 6, 12, 18, 24, 27, 33, 36, 39, 42, 48, 51, 54 and 60 months in the following QoL scales: Fatigue, Physical Functioning and Global Health Status/QoL (outcome measure: EORTC QLQ-C30), Impact on Daily Life and Symptom Burden (outcome measure: EORTC CML-24), Burden of Illness (outcome measure: EORTC QLQ-ELD14).

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Pane, Study Chair — Università Federico II of Naples
Locations (82):
- Italy (76):
  - S.O.C. di Ematologia - Azienda Ospedaliera - SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Azienda Ospedaliero - Universitaria Ospedali Riuniti Umberto I - G.M. Lancisi G. Salesi, Ancona
  - Area Vasta N. 5 Ascoli Piceno - S. Benedetto Del Tronto, Presidio Ospedaliero Av5 Osp. Gen. Prov.Le "C.G.Mazzoni" - Uoc Ematologia, Ascoli Piceno
  - Asl Di Asti, Ospedali Riuniti - Presidio Ospedaliero Cardinal G. Massaia - Sc Oncologia, Asti
  - Ao Di Rilievo Nazionale E Di Alta Specialità "San Giuseppe Moscati" - Avellino - Uoc Ematologia Con Unità Di Trapianto, Avellino
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - Asl Della Provincia Di Barletta, Andria, Trani, Ospedale "Mons. Dimiccoli" - Barletta - Uo Ematologia, Barletta
  - Ematologia Torre 6 piano 4 - ASST Papa Giovanni XXIII, Bergamo
  - Istituto di Ematologia "Lorenzo e A. Seragnoli" - Università degli Studi di Bologna - Policlinico S. Orsola - Malpighi, Bologna
  - USD Trapianti di midollo per adulti - Cattedra di Ematologia - Università degli Studi di Brescia, Brescia
  - ASL N.8 -Ospedale A. Businco, Cagliari
  - Cagliari CTMO - Ematologia - Ospedale "Binaghi", Cagliari
  - Gemelli Molise - Campobasso - Uosd Onco-Ematologia, Campobasso
  - U.O.C. Oncoematologia - Istituto Oncologico Veneto Irccs, Presidio Ospedaliero S. Giacomo Apostolo, Castelfranco Veneto
  - Università di Catania - Cattedra di Ematologia - Ospedale "Ferrarotto", Catania
  - Ao Di Catanzaro "Pugliese-Ciaccio", Presidio Ospedaliero "Ciaccio - de Lellis" - Ematologia, Catanzaro
  - U.O. di Medicina Interna - ASUR Marche 8 - Ospedale Civile, Civitanova Marche
  - Azienda Ospedaliero Universitaria Arcispedale Sant'Anna Dipartimento di Scienze Mediche Sezione di Ematologia e Fisiopatologia dell'Emostasi, Cona
  - Ao Di Cosenza, Presidio Ospedaliero Annunziata - Uoc Ematologia, Cosenza
  - S.C. Ematologia ASO S. Croce e Carle, Cuneo
  - Unità di Ricerca e di Malattie del sangue - Ematologia San Luca Vecchio Pad. 16 - 1° Piano, Florence
  - Aou Ospedali Riuniti - Foggia - Uoc Ematologia, Foggia
  - Irccs Aou San Martino - Genova - Uo Ematologia E Trapianti, Genova
  - IRCCS_AOU San Martino-IST.Clinica Ematologica, Genova
  - Asl Latina, Presidio Ospedaliero Nord - Ospedale Santa Maria Goretti - Uoc Ematologia, Latina
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - I.R.S.T. Srl Irccs - Meldola - Sc Oncologia Medica, Meldola
  - Azienda Ospedaliera Universitaria - Policlinico G. Martino Dipartimento di Medicina Interna - U.O. Messina, Messina
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - U.O. di Ematologia- Ospedale dell'Angelo - Mestre, Mestre
  - Fondazione Irccs "Istituto Nazionale Tumori" - Milano - Sc Ematologia, Milan
  - Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico - Milano - Ematologia - Padiglione Marcora, Milan
  - UO Ematologia - AOU Policlinico di Modena, Modena
  - Asl Napoli 1 Centro, Presidio Ospedaliero Ascalesi - Ospedale S.Maria Di Loreto Nuovo, Napoli
  - Azienda Ospedaliera di Rilievo Nazionale A. Cardarelli, Napoli
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - Ospedale San Gennaro - ASL Napoli 1, Napoli
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - U.O. CTMO Ematologia - Osp. S. Francesco, Nuoro
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga-Medicina Interna 2, Orbassano
  - Aou Di Padova - Uo Ematologia, Padua
  - Asl Salerno, Presidio Ospedaliero Tortora Pagani - Ematologia, Pagani
  - Ospedali Riuniti "Villa Sofia-Cervello", Palermo
  - U.O. di Ematologia con trapianto - Centro di Riferimento Regionale per le coagulopatie rare nel bambino e nell'adulto Dipart. Biomedico di Medicina Interna - A.U. Policlinico "Paolo Giaccone", Palermo
  - Aou Di Parma - Sc Ematologia E Centro Trapianti Midollo Osseo, Parma
  - Div. di Ematologia di Muraglia - CTMO Ospedale San Salvatore, Pesaro
  - Asl Pescara, Presidio Ospedaliero 'Spirito Santo' - Uoc Ematologia Clinica, Pescara
  - Unità Operativa Ematologia e Centro Trapianti - Dipartimento di Oncologia ed Ematologia - AUSL Ospedale G. da Saliceto, Piacenza
  - Az.Ospedaliera S.G.Moscati, Potenza
  - Dipartimento Oncologico - Ospedale S.Maria delle Croci, Ravenna
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - Unità Operativa Complessa di Ematologia - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ausl Della Romagna, Ospedale "Infermi" - Rimini - Uo Ematologia, Rimini
  - Asl Roma 2, Ospedale S. Eugenio- Ospedale S.Eugenio - Uoc Ematologia, Roma
  - Az. Ospedaliera "Sant' Andrea"-Università la Sapienza Seconda Facoltà di Medicina e Chirurgia, Roma
  - Divisione Ematologia - Università Campus Bio-Medico, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - UOC Pronto Soccorso e Accettazione Ematologica - Dipartimento Biotecnologie Cellulari ed Ematologia - Università degli Studi di Roma "Sapienza", Roma
  - U.O.C. Ematologia - Ospedale S. Eugenio, Rome
  - Unità Operativa di Oncologia Giovanni Paolo II "Vito Fazzi", Rossano
  - Aulss 5 Polesana, Presidio Ospedaliero Di Rovigo - Uosd Ematologia, Rovigo
  - Aou "San Giovanni Di Dio E Ruggi D'Aragona" - Salerno - Uoc Ematologia E Trapianti Di Cellule Staminali Emopoietiche, Salerno
  - Istituto di Ematologia - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ematologia - Dipartimento di Medicina Clinica e Sperimentale, Sassari
  - Ospedale Di Sassuolo Spa - Ematologia, Sassuolo
  - Aou Senese - Uoc Ematologia E Trapianti, Siena
  - A.O. Santa Maria - Terni S.C Oncoematologia, Terni
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia - Università Degli Studi Di Torino, Torino
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia 2, Torino
  - Ospedale Mauriziano Umberto I - Torino - Scdu Ematologia, Torino
  - Unità Operativa Di Ematologia - Presidio Ospedaliero Di Treviso - Azienda Ulss N.2 Marca Trevigiana, Treviso
  - Clinica Ematologica-Centro Trapianti e Terapie cellulari Azienda Ospedaliero-Universitaria, Udine, Udine
  - Università degli Studi di Verona - A. O. - Istituti Ospitalieri di Verona- Div. di Ematologia - Policlinico G.B. Rossi, Verona
  - Aulss 8 Berica - Ospedale Di Vicenza - Uoc Ematologia, Vicenza
  - ULSS N.6 Osp. S. Bortolo, Vicenza
- Netherlands (6):
  - Meander Mc - Paesi Bassi, Amersfoort
  - Vumc - Paesi Bassi, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - A. Schweitzer Zh, Dordwijk - Paesi Bassi, Dordrecht
  - Zuyderland Medical Center - Paesi Bassi, Heerlen
  - Spaarne Ziekenhuis - Paesi Bassi, Hoofddorp

IPD SHARING:
Plan to Share IPD: No